CLINICAL TRIAL: NCT00071708
Title: Open Label Duloxetine Compassionate Use in Patients Who Have Completed a Previous Neuroscience Duloxetine Clinical Trial
Brief Title: Duloxetine Compassionate Use in Patients Who Have Completed a Previous Neuroscience Duloxetine Clinical Trial
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 7443; F1J-MC-HMCN
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Fibromyalgia; Diabetic Peripheral Neuropathic Pain; Generalized Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Fibromyalgia; Generalized Anxiety Disorder | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride

SUMMARY:
The primary objective of this study is to provide duloxetine to investigators for the treatment of patients who have previously participated in neuroscience duloxetine clinical trials and for whom effective alternative therapy is not available.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female outpatients at least 18 years of age who have previously participated in a Lilly sponsored neuroscience duloxetine clinical trial
* All females must have a negative urine pregnancy test at visit 1. Females of childbearing potential must agree to utilize medically acceptable and reliable means of birth control.
* Must sign the informed consent document

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug except for duloxetine that has not received regulatory approval for any indication at the time of study entry
* In the opinion of the investigator, patient judged to be at serious suicidal risk.
* Serious or unstable hepatic or renal function or unstable narrow angle glaucoma.
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to visit 1 or potential to use a MAOI during the study or within 5 days of discontinuation of study drug.
* Any patient who previously experienced a serious adverse event while taking duloxetine unless approved by the Lilly Physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Australia (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paddington, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everton Park, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maroochydore, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southport, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Hill, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoppers Crossing, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Perth, Western Australia

REFERENCES:
- [Derived] Pangallo BA, Zhang Q, Desaiah D, Perahia DG, Detke MJ, Kennedy SH. Long-term safety of duloxetine during open-label compassionate use treatment of patients who completed previous duloxetine clinical trials. Curr Med Res Opin. 2010 Nov;26(11):2643-51. doi: 10.1185/03007995.2010.522157. Epub 2010 Oct 11. PMID 20932222